CLINICAL TRIAL: NCT00124007
Title: A Phase I, Randomized, Placebo-Controlled, Double-Blind Trial to Evaluate the Safety and Immunogenicity of a Multiclade HIV-1 DNA Plasmid Vaccine Followed by Recombinant, Multiclade HIV-1 Adenoviral Vector Vaccine or the Multiclade HIV-1 Adenoviral Vector Vaccine Alone in Healthy Adult Volunteers Not Infected With HIV
Brief Title: Safety of and Immune Response to an Adenoviral HIV Vaccine (VRC-HIVADV014-00-VP) With or Without a Plasmid HIV Vaccine (VRC-HIVDNA016-00-VP) in HIV Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IAVI V001; 10380 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: VRC-HIVADV014-00-VP
Biological: VRC-HIVDNA016-00-VP

SUMMARY:
The purpose of this study is to determine the safety of and immune response to an investigational HIV vaccine, VRC-HIVADV014-00-VP, with or without a second investigational HIV vaccine, VRC-HIVDNA016-00-VP, in HIV uninfected adults.

DETAILED DESCRIPTION:
The worldwide HIV/AIDS epidemic may only be controlled through development of a safe and effective vaccine that will prevent HIV infection. This study will evaluate the safety and immunogenicity of an experimental adenovirus-vectored multiclade HIV vaccine, VRC-HIVADV014-00-VP, followed with either a similarly structured DNA plasmid HIV vaccine, VRC-HIVDNA016-00-VP, or a placebo. The DNA plasmids in both vaccines code for proteins from HIV subtypes A, B, and C, which together represent 90% of new HIV infections in the world. HIV uninfected volunteers will be recruited in Kenya and Rwanda.

Volunteers will participate in this study for 1 year. Participants will be randomly assigned to one of four groups:

* Group A participants will receive a low dose of the adenovirus-vectored vaccine or placebo at study entry.
* Group B participants will receive a higher dose of the adenovirus-vectored vaccine or placebo at study entry.
* Group C participants will receive the DNA plasmid vaccine or placebo at study entry and Months 1 and 2. They will receive either a low dose of the adenovirus-vectored vaccine or placebo at Month 6.
* Group D participants will receive the DNA plasmid vaccine or placebo at study entry and Months 1 and 2. They will receive either a higher dose of the adenovirus-vectored vaccine or placebo at Month 6.

All participants will undergo vital signs measurements before and after receiving each vaccination.

Participants in Groups A and B will have 9 study visits over 12 months. A physical exam, adverse events reporting, and medical and medication history will occur at each visit. HIV testing and counseling and blood and urine collection will occur at selected visits.

Participants in Groups C and D will have 17 study visits over 12 months. A physical exam, adverse events reporting, and medical and medication history will occur at each visit. HIV testing and counseling and blood and urine collection will occur at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* Willing to follow all the requirements of the study and available for follow-up for the duration of the study
* Have understanding of the study and provide written informed consent
* Willing to undergo HIV testing and counseling and willing to receive HIV test results
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* HIV infected
* Hepatitis B virus infected
* Hepatitis C virus infected
* Active or untreated syphilis
* Participated in high-risk behavior for HIV infection within 6 months prior to study entry. More information on this criterion can be found in the protocol.
* Any clinically significant abnormality in history or upon examination (e.g., immunodeficiency or autoimmune disease; use of systemic corticosteroids, immunosuppressive, antiviral, anticancer, or other medications considered significant by the investigator) within 6 months prior to study entry
* Any clinically significant acute or chronic medical condition that, in the opinion of the investigator, would make the volunteer unsuitable for the study
* Live attenuated vaccines within 30 days prior to study entry OR plan to receive a live attenuated vaccine within 60 days after vaccination in this study
* Subunit or killed vaccines within 14 days prior to study entry OR plan to receive a subunit or killed vaccine within 14 days after vaccination in this study
* Blood transfusion or blood products within 120 days prior to study entry
* Immunoglobulin within 60 days prior to study entry
* Participation in another investigational product clinical trial in the 3 months prior to study entry OR expected to participate in another investigational trial during this study
* Any other investigational HIV vaccine at any time
* History of severe local or systemic reactogenicity to vaccines or history of severe allergic reactions
* Major psychiatric illness, including any history of schizophrenia or severe psychosis, bipolar disorder requiring therapy, or suicide attempt or suicidal thoughts within the 3 years prior to study entry
* Uncontrolled hypertension
* Pregnant, breastfeeding, or plan to become pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2005-11; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Local reactogenicity signs and symptoms
systemic reactogenicity signs and symptoms
laboratory measures of safety
adverse and serious adverse experiences

SECONDARY OUTCOMES:
Proportion of volunteers who have HIV-1 specific T-cell responses quantified by intracellular cytokine staining (ICS; both CD4+ and CD8+) and ELISPOT and magnitude of the responses
proportion of volunteers with HIV-1 specific antibodies and magnitude of the response
proportion of volunteers with increase in antibodies to rAd5
impact of pre-existing immunity to rAd5 on immunogenicity
proportion of volunteers who test "false positive" on standard HIV testing algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Job Bwayo, MD, PhD, Principal Investigator — Kenya AIDS Vaccine Initiative, University of Nairobi; Etienne Karita, MD, Principal Investigator — Project San Francisco
Locations (3):
- Kenya (2):
  - KEMRI, Ctr. for Geographic Medicine Research Coast at Kilifi, Kilifi
  - KAVI, KNH at Kangemi, Nairobi
- Projet San Francisco, Kigali, Rwanda

REFERENCES:
- [Background] Esparza J, Osmanov S. HIV vaccines: a global perspective. Curr Mol Med. 2003 May;3(3):183-93. doi: 10.2174/1566524033479825. PMID 12699356
- [Background] Gaschen B, Taylor J, Yusim K, Foley B, Gao F, Lang D, Novitsky V, Haynes B, Hahn BH, Bhattacharya T, Korber B. Diversity considerations in HIV-1 vaccine selection. Science. 2002 Jun 28;296(5577):2354-60. doi: 10.1126/science.1070441. PMID 12089434
- [Background] Stratov I, DeRose R, Purcell DF, Kent SJ. Vaccines and vaccine strategies against HIV. Curr Drug Targets. 2004 Jan;5(1):71-88. doi: 10.2174/1389450043490686. PMID 14738219
- [Derived] Omosa-Manyonyi GS, Jaoko W, Anzala O, Ogutu H, Wakasiaka S, Malogo R, Nyange J, Njuguna P, Ndinya-Achola J, Bhatt K, Farah B, Oyaro M, Schmidt C, Priddy F, Fast P. Reasons for ineligibility in phase 1 and 2A HIV vaccine clinical trials at Kenya AIDS vaccine initiative (KAVI), Kenya. PLoS One. 2011 Jan 21;6(1):e14580. doi: 10.1371/journal.pone.0014580. PMID 21283743
- [Derived] Jaoko W, Karita E, Kayitenkore K, Omosa-Manyonyi G, Allen S, Than S, Adams EM, Graham BS, Koup RA, Bailer RT, Smith C, Dally L, Farah B, Anzala O, Muvunyi CM, Bizimana J, Tarragona-Fiol T, Bergin PJ, Hayes P, Ho M, Loughran K, Komaroff W, Stevens G, Thomson H, Boaz MJ, Cox JH, Schmidt C, Gilmour J, Nabel GJ, Fast P, Bwayo J. Safety and immunogenicity study of Multiclade HIV-1 adenoviral vector vaccine alone or as boost following a multiclade HIV-1 DNA vaccine in Africa. PLoS One. 2010 Sep 21;5(9):e12873. doi: 10.1371/journal.pone.0012873. PMID 20877623